CLINICAL TRIAL: NCT02636387
Title: Desmopressin as a Therapy for Nocturnal Enuresis in Patients With Sickle Cell Disease
Brief Title: Desmopressin as a Therapy for Bedwetting in Children With Sickle Cell Disease
Status: Terminated | Type: Observational
Why Stopped: Low recruitment
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Kerry Morrone, Assistant Professor of Pediatrics, Montefiore Medical Center
Other Study IDs: 2014-3768
Record Dates: First submitted 2015-12-17; First posted 2015-12-21 (Estimated); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Nocturnal Enuresis; Anemia, Sickle Cell
MeSH Terms: conditions — Nocturnal Enuresis; Anemia, Sickle Cell | interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Desmopressin: 0.2mg tablets, dose titrated to effect
  Interventions: Drug: Desmopressin
- Placebo: Placebo Comparator

INTERVENTIONS:
Drug: Desmopressin — Two desmopressin 0.2 mg tablets at bedtime for 14 days and monitoring if <50 % improvement
  Other Names: DDAVP
  Groups: Desmopressin

SUMMARY:
This study assesses if using the medication desmopressin will decrease nightime bedwetting in children with sickle cell disease.

DETAILED DESCRIPTION:
Night time bedwetting is a common complication of sickle cell disease, and affects up to 30 % of children . Desmopressin is an oral medication that increases water reabsorption in the kidneys. Studies have shown that it is effective in decreasing bedwetting episodes in children without sickle cell disease. Chronic sickling episodes causing damage to the kidneys could cause permanent damage and may make this treatment ineffective in sickle cell disease. This trial will inform pediatric sickle cell doctors if desmopressin is an appropriate treatment for bed wetting in the investigators patients.

This work is being continued on study ID: 2020-11268.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Hemoglobin SS, SC, SB0thal or SB+thal
2. Patients with at least two episodes of primary nocturnal enuresis per week or four episodes over the two weeks prior to enrollment.
3. Patients with secondary enuresis who have been evaluated and cleared by a pediatric urologist as not having other etiologies of enuresis (e.g. overactive detrusor activity, a genitourinary anatomic abnormality)

Exclusion Criteria:

1. Patients with developmental delay or neurologic dysfunction secondary to stroke.
2. Patients with hypertension or underlying renal disease.
3. Patients with genitourinary anatomic abnormalities. Any prior renal ultrasound showing normal genitourinary anatomy is sufficient to clear a patient for the study.
4. Patients with daytime urinary incontinence
5. Patients with glucosuria on urinalysis.
6. Patients with secondary nocturnal enuresis who have not been evaluated by a pediatric urologist to rule out other etiologies of enuresis.
7. Patients who are pregnant.
8. Patients receiving another medicine for nocturnal enuresis (e.g. imipramine).

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will consist of children (ages 8-21) with Hemoglobin SS, SC, SB0thal or SB+thal and with Nocturnal Enuresis who are treated at the children's hospitals outpatient hematology clinic and/or the inpatient hematology unit.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2015-08-26 (Actual); Primary Completion 2018-10-27 (Actual); Study Completion 2018-10-27 (Actual)

PRIMARY OUTCOMES:
Reduction in Bedwetting episodes | Baseline and 4 weeks
  To prospectively assess if the use of desmopressin in patients with sickle cell disease and nocturnal enuresis will decrease the number of nighttime episodes of enuresis by 50% after initiating DDAVP at 0.4 mg nightly dose with dose escalation as clinically indicated compared to the control group.

SECONDARY OUTCOMES:
Quality of life measure | Baseline and 4 weeks
  To determine if patients with sickle cell disease and nocturnal enuresis receiving desmopressin will have an improved quality of life compared to the control group.
Reduction in Nighttime awakenings | Baseline and 4 weeks
  To determine if the use of desmopressin in patients with nocturnal enuresis improves rates of nocturia, defined as episodes of nighttime awakening to void in children ≥5 years of age, compared to the control group.
Reduction in Daytime Fatigue | Baseline and 4 weeks
  To determine if patients with sickle cell disease and nocturnal enuresis receiving desmopressin will have less daytime fatigue compared to the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Kerry A Morrone, MD, Principal Investigator — Children's Hospital at Montefiore
Locations (1):
- Children's Hospital at Montefiore, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neveus T, von Gontard A, Hoebeke P, Hjalmas K, Bauer S, Bower W, Jorgensen TM, Rittig S, Walle JV, Yeung CK, Djurhuus JC. The standardization of terminology of lower urinary tract function in children and adolescents: report from the Standardisation Committee of the International Children's Continence Society. J Urol. 2006 Jul;176(1):314-24. doi: 10.1016/S0022-5347(06)00305-3. PMID 16753432
- [Background] Barakat LP, Smith-Whitley K, Schulman S, Rosenberg D, Puri R, Ohene-Frempong K. Nocturnal enuresis in pediatric sickle cell disease. J Dev Behav Pediatr. 2001 Oct;22(5):300-5. doi: 10.1097/00004703-200110000-00004. PMID 11718233
- [Background] Readett DR, Morris JS, Serjeant GR. Nocturnal enuresis in sickle cell haemoglobinopathies. Arch Dis Child. 1990 Mar;65(3):290-3. doi: 10.1136/adc.65.3.290. PMID 2334206
- [Background] Field JJ, Austin PF, An P, Yan Y, DeBaun MR. Enuresis is a common and persistent problem among children and young adults with sickle cell anemia. Urology. 2008 Jul;72(1):81-4. doi: 10.1016/j.urology.2008.02.006. Epub 2008 Apr 2. PMID 18384865
- [Background] Naitoh Y, Kawauchi A, Soh J, Kamoi K, Miki T. Health related quality of life for monosymptomatic enuretic children and their mothers. J Urol. 2012 Nov;188(5):1910-4. doi: 10.1016/j.juro.2012.07.012. Epub 2012 Sep 19. PMID 22999692
- [Background] Glazener CM, Evans JH. Desmopressin for nocturnal enuresis in children. Cochrane Database Syst Rev. 2002;(3):CD002112. doi: 10.1002/14651858.CD002112. PMID 12137645
- [Background] Becker AM. Sickle cell nephropathy: challenging the conventional wisdom. Pediatr Nephrol. 2011 Dec;26(12):2099-109. doi: 10.1007/s00467-010-1736-2. Epub 2011 Jan 4. PMID 21203778
- [Background] Statius van Eps LW, Schouten H, Haar Romeny-Wachter CC, La Porte-Wijsman LW. The relation between age and renal concentrating capacity in sickle cell disease and hemoglobin C disease. Clin Chim Acta. 1970 Mar;27(3):501-11. doi: 10.1016/0009-8981(70)90305-0. No abstract available. PMID 5435231
- [Background] Figueroa TE, Benaim E, Griggs ST, Hvizdala EV. Enuresis in sickle cell disease. J Urol. 1995 Jun;153(6):1987-9. PMID 7752379
- [Background] Robson WL, Leung AK, Norgaard JP. The comparative safety of oral versus intranasal desmopressin for the treatment of children with nocturnal enuresis. J Urol. 2007 Jul;178(1):24-30. doi: 10.1016/j.juro.2007.03.015. Epub 2007 May 11. PMID 17574054